CLINICAL TRIAL: NCT00031798
Title: A Phase III, Double-Blind, Prospective Randomized Clinical Trial of the Effect of D-threo-methylphenidate HCl (d-MPH) on Quality of Life in Brain Tumor Patients Receiving Radiation Therapy
Brief Title: Methylphenidate to Improve Quality of Life in Patients Undergoing Radiation Therapy for Brain Tumors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual; loss of funding
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: REBACDR0000069227; CCCWFU-97600; NCI-P02-0211
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Depression; Fatigue; Quality of Life
Keywords: fatigue; depression; quality of life; cognitive/functional effects; recurrent adult brain tumor; adult brain stem glioma; adult glioblastoma; adult tumors metastatic to brain; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult meningioma; adult anaplastic ependymoma; adult myxopapillary ependymoma; adult ependymoblastoma; adult pilocytic astrocytoma; adult subependymoma; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma; adult grade II meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Depression; Fatigue; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Meningioma; Ependymoma; Neuroectodermal Tumors, Primitive; Glioma, Subependymal; Gliosarcoma | interventions — Methylphenidate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: methylphenidate hydrochloride
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Methylphenidate may decrease side effects of radiation therapy. It is not yet known if methylphenidate is effective in improving quality of life in patients with primary or metastatic brain tumors.

PURPOSE: Randomized phase III trial to determine the effectiveness of methylphenidate in improving quality of life in patients who have brain tumors and are undergoing radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of d-methylphenidate on fatigue in patients receiving radiotherapy for primary or metastatic brain tumors.
* Determine the effect of this drug on the quality of life of these patients.
* Determine the effect of this drug on depression in these patients.
* Determine the effect of this drug on global neurocognitive function, including attention and concentration, memory, language, visuospatial skills, and executive function, in these patients.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified by tumor type (primary vs metastatic), treatment (radiotherapy vs radiotherapy and chemotherapy), and Karnofsky performance status (70% or 80% vs 90% or 100%). Patients are randomized to one of two treatment arms.

All patients undergo radiotherapy over weeks 1-4.

* Arm I: Patients receive oral d-methylphenidate twice daily on weeks 1-12.
* Arm II: Patients receive oral placebo twice daily on weeks 1-12. In both arms, quality of life is assessed at baseline, at the end of radiotherapy, and at 4, 8, and 12 weeks after radiotherapy.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 200 patients (100 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic brain tumor OR
* Histologically confirmed primary brain tumor

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Low-grade glioma
  * Meningioma
  * Ependymoma
* Planned external beam cranial radiotherapy (partial or whole brain) with a total dose of at least 25 Gy in at least 10 fractions of 180-300 cGy each

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC ≥ 1,500/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥ 75,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No hypertension or other cardiovascular disease requiring antihypertensives and/or other cardiovascular medications

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious medical or psychiatric illness that would preclude study participation
* No hypersensitivity to study drug
* No history of steroid psychosis
* No family history of or active Tourette's Syndrome
* No prior or active glaucoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior or concurrent chemotherapy allowed

Endocrine therapy:

* Concurrent steroids allowed

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy allowed except to brain (including stereotactic radiosurgery)
* No concurrent craniospinal axis radiotherapy

Surgery:

* Not specified

Other:

* No prior or concurrent medications for attention deficit disorder, anxiety disorder, schizophrenia, or substance abuse
* No concurrent anti-depressants

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04-01 (Actual); Primary Completion 2005-03-01 (Actual); Study Completion 2006-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Central Illinois, Decatur, Illinois
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Upstate Carolina, Spartanburg, South Carolina